CLINICAL TRIAL: NCT03019562
Title: Oxycodone vs. Fentanyl in the Treatment of Early Postoperative Pain After Total Hip Replacement
Brief Title: Oxycodone vs. Fentanyl in Early Postoperative Pain After Total Hip Replacement
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Mi Kyeong Kim, Associate Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KHUH 2016-09-047
Record Dates: First submitted 2017-01-11; First posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Pain, Postoperative
Keywords: postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Oxycodone; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxycodone (Experimental): 4mg of oxycodone iv bolus
  Interventions: Drug: Oxycodone
- Fentanyl (Active Comparator): 50ug of fentanyl iv bolus
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Oxycodone — 4mg of oxycodone iv 20 min before the end of surgery, 10ug/kg of fentanyl in Patient-Controlled Analgesia(PCA)
  Other Names: Oxynorm
  Arms: Oxycodone
Drug: Fentanyl — 50ug of fentanyl iv 20 min before the end of surgery, 10ug/kg of fentanyl in Patient-Controlled Analgesia(PCA),
  Arms: Fentanyl

SUMMARY:
Oxycodone is one of the most widely used opioids for pain treatment. Many studies demonstrated good efficacy of oxycodone on postoperative pain. In this study, we assess the efficacy and side effects of bolus intravenous of oxycodone injection compared to those of fentanyl in patients after total hip replacement surgery.

DETAILED DESCRIPTION:
Oxycodone is one of the most widely used opioids for pain treatment. There have been several studies on the efficacy and side effects of oxycodone. Oxycodone has been known to have the same potency with morphine. Many studies demonstrated good efficacy of oxycodone on postoperative pain. In this study, we designed a prospective, randomized, and double-blind study to assess the efficacy and side effects of bolus intravenous of oxycodone injection compared to those of fentanyl in patients who underwent the total hip replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* 19-65 years of age
* ASA physical status classification I or II
* Scheduled for total hip replacement surgery

Exclusion Criteria:

* Allergic to study drugs
* Patient with asthma or COPD, patient who is severely respiratory depressed
* Renal of hepatic insufficiency
* Epileptic status
* Intracranial lesion associated with increased intracranial pressure
* Acute abdomen, patient who has diagnosed paralytic ileus or suspicious ileus
* Pregnant or lactating women

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain measurement using Numeric Rating Scale(NRS) | Immediately after surgery
  Measure postoperative pain using NRS at the PostAnesthesia Care Unit(PACU)

SECONDARY OUTCOMES:
Additional doses of fentanyl for pain management | From immediately after surgery to 2 days after surgery
  0-6 hours, 6-12 hours, 12-24 hours, 24-48 hours after surgery

OTHER OUTCOMES:
Adverse effect | From immediately after surgery to 2 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mi Kyeong Kim, MD, PhD, Principal Investigator — Kyunghee University Medical Center
Locations (1):
- Kyung Hee University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No